CLINICAL TRIAL: NCT02214173
Title: The Effect of an Enhanced Rice Bran Nutritional Supplement on Metabolic Syndrome Variables in HIV
Brief Title: The Effect of an Enhanced Rice Bran Nutritional Supplement in HIV
Acronym: BRM4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Daiwa Health Development (Other)
Responsible Party: Principal Investigator, John E. Lewis, Principal Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20130279
Record Dates: First submitted 2014-08-01; First posted 2014-08-12 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: HIV, BRM4, hydrolyzed rice bran, metabolic syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rice bran arabinoxylan compound (RBAC) (Experimental): 2 capsules with 6 to 8 ounces of water 3 times per day (6 tablets total per day) for 6 months.
  Interventions: Dietary Supplement: rice bran arabinoxylan compound (RBAC)
- placebo (Placebo Comparator): 2 capsules with 6 to 8 ounces of water 3 times per day (6 tablets total per day) for 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: rice bran arabinoxylan compound (RBAC) — 2 capsules with 6 to 8 ounces of water 3 times per day (6 tablets total per day) for 6 months.
  Arms: rice bran arabinoxylan compound (RBAC)
Dietary Supplement: Placebo — 2 capsules with 6 to 8 ounces of water 3 times per day (6 tablets total per day) for 6 months.
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effects of the nutritional supplement rice bran arabinoxylan compound (RBAC) on metabolic syndrome variables in persons living with HIV. The hypothesis is that there will be a significant improvement in metabolic syndrome and immune variables in HIV-positive participants in the intervention group compared to the control group.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of Rice Bran Arabinoxylan Compound (RBAC) on metabolic syndrome variables in persons living with HIV (PLWH). This nutritional supplement is made from a water soluble extract of rice bran that has been partially hydrolyzed by the action of a natural enzyme complex extracted from Shiitake mushroom. Given that these micronutrients may be important for regulating the immune system and metabolizing glucose, the investigators will explore the impact of RBAC on metabolic syndrome (MetSyn) variables according to the National Cholesterol Education Program (NCEP) Adult Treatment Panel III guidelines (1) (fasting plasma glucose, waist circumference, high-density lipoprotein [HDL] cholesterol, triglycerides, and blood pressure), secondarily on additional atherogenic variables (total cholesterol, low-density lipoprotein [LDL] cholesterol, hip circumference, and body mass index) and immune functioning (CD4+ and CD8+) among 40 HIV+ adult (18+ years of age and over) patients on stable antiretroviral therapy (ART). Specifically, subjects will participate in a 6-month, two-group, randomized intervention, where one group (n=20) will take 3 gram/day RBAC and the other group (n=20) will take a placebo to compare differences in outcomes between the two groups. The results of the study are intended to address the multi-faceted physiological problems of HIV+ patients by testing the efficacy of a nutritional supplement intervention on multiple outcomes in this population.

No substantial psychological, medical, or social risks exist to the participants, other than minor discomfort associated with the venipuncture. Although all measures to protect confidentiality will be put in place, the possibility exists that electronic data could be jeopardized. In the remote case that such event occurs, it will be immediately reported to the Institutional Review Board.

The components of RBAC should be harmless without significant food allergies. No serious, untoward side effects have been reported to the company by consumers nor observed during previous human studies. Potential adverse effects will be explained to each participant when informed consent is obtained. Whole foods supplements are virtually no different than consuming food, because of how they are manufactured. The investigators prior study on RBAC showed no adverse effects. If any side effect does occur, the remedy is to discontinue until asymptomatic, and then reintroduce at 1/4 dosage, increasing by the same amount every 2 days, if uneventful, until full dosage is achieved. Study staff will provide additional follow-up and consultation with any subject who experiences an untoward side effect.

Other potential risks include:

1. Randomization. A potential risk for the placebo group is no improvement in the investigators outcomes of interest.
2. Data collection. The investigators foresee minimal risks associated with the testing, other than discomfort or fatigue.

A toxicology search for each component reveals no unique toxicity characteristic of the materials. As reported by Daiwa Health Development, the manufacturer of the product, thousands of people currently use RBAC (under the trade names BRM4 and PeakImmune 4), and Daiwa is unaware of significant toxicities. Daiwa applies the latest scientific methods to ensure the value and safety of their raw materials. Daiwa products are manufactured in state-of-the-art facilities, under strict quality control and environmental protection standards.

Participants will incur no additional appreciable psychological or social risks by participating in this study, although they may undergo psychological and physical discomfort sometimes. The process of interviewing during the assessment may cause discomfort. Discomfort or fatigue may also be experienced in completing the assessment battery.

Alternatives to this study for these MetSyn and immune functioning variables include prescription medications, exercise, dietary modification, and other nutritional supplements. The risks of medications can be very significant, including life-threatening, but the risk of taking nutritional supplements is not totally understood, since they are not regulated by the US Food and Drug Administration. Medications and nutritional supplements, as part of a change in lifestyle behaviors, may also prove to be beneficial for MetSyn variables and immune system functioning, but their long-term use has unknown consequences.

The information obtained in this study will help in determining the efficacy of using RBAC on MetSyn and metabolic variables and immune system functioning. By participating in the study, subjects may experience improved health status. The risk of participating in this study is reasonable because of the potential enhancements in metabolic and immune system functioning with improved nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Confirmed HIV infection
3. CD4 T cell counts > 50/µl and < 250/µl
4. On a stable ART regimen (e.g., Kaletra-based) before (≤6 months) and during the intervention
5. Planning to maintain current medication during the course of the intervention
6. Not on any lipid-lowering agents for a minimum of 3 months before the enrollment
7. Previous nutritional supplement usage of similar polysaccharide formula permitted, but current use must be stopped 2 weeks before and during trial
8. Interested in participating in a dietary supplement study
9. Willing to follow recommendations for participating in the study
10. Willing to not consume food, alcohol, caffeine, or stimulants (amphetamines) 12 hours before each assessment
11. Able to provide informed consent

Exclusion Criteria:

1. Currently enrolled in another research trial for similar investigative nutritional therapies
2. Known allergy to rice, rice bran, mushrooms, or related food products
3. Any gastrointestinal disorders that could lead to uncertain resorption of the study supplement
4. Other medical complications that might preclude one from participating in the study, i.e., recent heart attack or stroke or chronic kidney disease
5. Currently taking immunomodulatory medication, i.e., interferon
6. Currently taking chemotherapeutic agents
7. Multiple drug resistance
8. Current smoker
9. Severe anemia or other medical condition that will not permit a safe blood draw
10. A bleeding disorder
11. A terminal illness
12. Women who are pregnant or are attempting conception, especially in the presence of a history of recurrent spontaneous abortion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Improvement in Metabolic Syndrome Markers | 3 months and 6 months
  Improvement in glucose, lipid profile, blood pressure, cluster of differentiation 4 (CD4), and cluster of differentiation 8 (CD8) values.

CONTACTS AND LOCATIONS:
Overall Officials: John E Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Clinical Research Building, Department of Psychiatry & Behavioral Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No